CLINICAL TRIAL: NCT03592147
Title: Identification of the Most Effective Relaxation Tool for Use in a Trial to Improve Breastfeeding Outcomes in Mothers of Late Preterm Infants: a Pilot Study
Brief Title: Investigation of Different Relaxation Techniques in Eliciting a Relaxation Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12521/001
Record Dates: First submitted 2018-07-05; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Stress, Psychological
Keywords: Meditation; Music; Relaxation; Light Therapy; Stress
MeSH Terms: conditions — Stress, Psychological | interventions — Mediation Analysis; Music Therapy; Meditation

STUDY DESIGN:
Intervention Model Description: Within-subject pilot study, where each participant will undergo five different relaxation therapies (guided imagery meditation, music listening, "relaxation" lighting, combination of light and meditation, and a combination of light and music) and one silence/control state.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Relaxation (Other): This is a within-subject pilot study, where each participant received, in random order, five different relaxation therapies (Guided Imagery Relaxation Tape, Music Listening, Relaxation Lighting, Meditation and Relaxation Light, and Music and Relaxation Light) and one Control/Silence state spanning across 3-6 weeks.
  Interventions: Other: Guided Imagery Relaxation Tape; Other: Music Listening; Other: Relaxation Lighting; Other: Meditation and Relaxation Light; Other: Music and Relaxation Light; Other: Control/Silence

INTERVENTIONS:
Other: Guided Imagery Relaxation Tape — The meditation is approximately 7 minutes in duration.
  Other Names: Mediation
Other: Music Listening — Participants have the option of selecting one of the following music categories: New age, classical, and oriental. The songs were selected based on criteria established in a previous study to induce relaxation. All songs were also modified in length to be approximately 7 minutes in duration.
  Other Names: Music
Other: Relaxation Lighting — The participants were asked to select either orange or blue lighting settings using the Philips Hue lighting. The intensity of the light will be fixed to control for that measure. They were asked to sit for approximately 7 minutes in duration.
Other: Meditation and Relaxation Light — The guided imagery meditation and relaxation lighting were combined.
Other: Music and Relaxation Light — The music and relaxation lighting were combined.
Other: Control/Silence — The participants were asked to relax for a duration of 7 minutes, with no explicit advice given. Lighting was adjusted to a specific intensity and colour (basic yellow light) as was used in the music and guided imagery interventions.

SUMMARY:
While the stress response, characterised by an increase in heart rate, blood pressure, and cortisol, has evolved to ensure the survival of the organism in face of danger, chronic stress due to psychological stressors can be harmful. The opposite of the stress response is the "relaxation response". Mind-body techniques such as meditation, guided imagery and music therapy are thought to induce this response. The relaxation response is characterized as a wakeful hypometabolic state, where a decrease in central nervous system arousal is observed. Some studies reported a reduction in stress hormones, and in symptoms of anxiety and depression following the use of mind-body relaxation techniques. Other studies noted a reduction in stress measured using physiological measurements such as heart rate and blood pressure.

Light therapy is another technique that is suggested to induce physiological changes similar to those seen in the relaxation response. Some studies have shown a reduction in heart rate, blood pressure, oxygen consumption and carbon dioxide production following exposure to blue light.

These relaxation therapies can be useful for the general population and for vulnerable groups where alternative therapies, such as medication and psychotherapy, are difficult. Limited amount of studies have quantified the decrease in stress in physiological measurements such as heart rate and blood pressure.

The aim of this study is to investigate which relaxation technique among five different interventions (and one control) is the most effective in improving relaxation and reducing stress in adult women of reproductive age (18-45 years). The results of this study will be used to inform the intervention of a study testing the impact of relaxation therapy on breastfeeding outcomes in mothers of late preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Women of reproductive age (18-45 years)
* Fluent in English

Exclusion Criteria:

* Any condition that may affect blood pressure, heart rate or energy expenditure i.e hypertension, hyperthyroidism, heart failure
* Smokers
* Recent surgeries or injuries

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-06-04 (Actual)

PRIMARY OUTCOMES:
Perceived Relaxation | Post-intervention, an average of 10 mins
  Perceived relaxation was assessed using a visual analogue scale (VAS), which is a 10 cm horizontal line spanning from the minimum to the maximum of the variable measured. The minimum (left) represents "completely unrelaxed" and the maximum (right) "completely relaxed". The women mark a point on the scale to indicate their feelings of relaxation. The distance between the mark and the minimum point was measured in centimetres (two decimal points).
Blood Pressure | Post-intervention, an average of 10 mins
  Systolic and diastolic blood pressure (mmHg) were measured three times using a digital sphygmomanometer.
Heart Rate | Post-intervention, an average of 10 mins
  Heart rate (bpm) was measured three times using a digital sphygmomanometer.
Fingertip Temperature | Post-intervention, an average of 10 mins
  A non-contact digital thermometer was used to measure fingertip temperature as an indication of sympathetic nervous system activation.

SECONDARY OUTCOMES:
Preference | At the end of the study, at approximately 3-6 weeks
  The women were asked to rank the relaxation therapies in order of preference

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Great Ormond Street Institute of Child Health, London, United Kingdom